CLINICAL TRIAL: NCT06312163
Title: Validation of Innovative Scheimpflug Topography Derived RGP Contact Lens Designs In Optometry Network
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: EHRD1001
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Keratoconus
Keywords: rigid gas permeable contact lens
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARM1: The contact lens to be investigated in this study (Scheimpflug topography derived corneal RGP contact lens design)
  Interventions: Device: The contact lens to be investigated in this study (Scheimpflug topography derived corneal RGP contact lens design). A CE (UKCA) marked class 2 medical devices.
- Arm2: The patient's own corneal RGP lens - CE (UKCA) marked class 2 medical devices.
  Interventions: Device: The contact lens to be investigated in this study (Scheimpflug topography derived corneal RGP contact lens design). A CE (UKCA) marked class 2 medical devices.

INTERVENTIONS:
Device: The contact lens to be investigated in this study (Scheimpflug topography derived corneal RGP contact lens design). A CE (UKCA) marked class 2 medical devices. — The participants will be fitted with (i) the optimal lens design as specified by the virtual fitting module, in addition to (ii) lenses that are one clinically significant step (0.12 mm) flatter and (iii) steeper in axial edge lift (AEL).

SUMMARY:
The goal of this Prospective, single-site, cohort study is to validate rigid gas permeable corneal contact lens (RGP) designs for keratoconus derived from combining the data from corneal topography scans and contact lenses ordered in patients with keratoconus (KC) attending a UK tertiary NHS Hospital contact lens clinic. The main questions it aims to answer are:

* Does a Scheimpflug topography derived RGP contact lens design for keratoconus have the equivalent overall contact lens fit as the patients' own lens?
* Is the number of trial lenses required to fit a patient is reduced compared to standard practice?
* Is the time taken to fit a contact lens is reduced compared to standard practice?
* Is there user acceptance of the new lens?
* Are the Axial ege lift (AEL) changes clinically significant?

There will be 3 work packages

WP1: For each participant data collection will take place over two visits.

• Visit 1: Pentacam topography scans and optimal 'virtual' lens selection will take place. • • Visit 2: Participants are fitted with 4 contact lenses (i) the optimal lens design as specified by the virtual fitting module, (ii) a contact lens with a clinically significant step flatter AEL (iii) a contact lens steeper in axial edge lift (AEL) (iv) the participant's own contact lens.

Each CL fit will be assessed with slit lamp photography according to the standardised method proposed by Wolffsohn et al. (2013), Anterior segment OCT MS39) (CSO Hansom Instruments, UK) and best-corrected visual acuity with each lens design using high-contrast logMAR .

WP2. Participants will attend one appointment where a traditional lens fit, and a lens fitted using the topography guided 'virtual' module will be undertaken (with the fitting method selected for each eye randomised). For each fitting method the total fitting time will be measured and the total number of trial contact lenses used. Patients will be invited to complete a questionnaire that probes their satisfaction of this process.

WP3. Clinicians not involved in the study will be invited to examine a demo version of the virtual fitting module and complete the validated system usability scale tool.

ELIGIBILITY:
Inclusion Criteria:

* - WP1:
* (a) Presence of keratoconus in either eye
* (b) Currently using a rigid gas permeable contact lens correction
* (c) Male or female, aged 18 years or older
* (d) The absence of significant media opacities
* (e) No ocular pathology other than keratoconus
* (f) Ability to understand nature/purpose of the study and to provide informed consent
* (g) Ability to follow instructions and complete the study
* (h) Ability to speak English
* WP2:
* (a) Presence of keratoconus in both eyes
* (b) Male or female, aged 18 years or older
* (c) The absence of significant media opacities
* (d) No ocular pathology other than keratoconus
* (e) Ability to understand nature/purpose of the study and to provide informed consent
* (f) Ability to follow instructions and complete the study
* (g) Ability to speak English
* WP3:
* (a) Optometrist, dispensing optician or ophthalmologist registered with the General Optical Council
* (b) Works within contact lens service at Moorfields Eye Hospital
* (c) Ability to understand nature/purpose of the study and to provide informed consent
* (d) Ability to follow instructions and complete the study
* (e) Ability to speak English .

Exclusion Criteria:

* - WP1:
* (a) Any systemic disease likely to affect visual performance
* (b) Any ocular disease that may affect visual performance, other than keratoconus
* (c) Hearing impairment sufficient to interfere with hearing instructions
* (d) Poor understanding of English language and/or alphabet
* (e) Any condition which, in the investigator's opinion, would conflict or otherwise prevent the participant from
* complying with the required procedures, schedule, or other study conduct.
* (f) Not currently using a rigid gas permeable contact lens or a contraindication to this
* (g) A history of corneal graft surgery (keratoplasty) in the eye under investigation.
* (h) A recent history (in preceding 12 months) of corneal abrasions in the designated study eye
* (i) A recent history (in preceding 1 month) of corneal cross linking for keratoconus
* WP2:
* (a) Any systemic disease likely to affect visual performance
* (b) Any ocular disease that may affect visual performance, other than keratoconus
* (c) Hearing impairment sufficient to interfere with hearing instructions
* (d) Poor understanding of English language and/or alphabet
* (e) Any condition which, in the investigator's opinion, would conflict or otherwise prevent the participant from
* complying with the required procedures, schedule, or other study conduct.
* (f) A contraindication to rigid gas permeable contact lens wear
* (g) A history of corneal graft surgery (keratoplasty) in the eye under investigation.
* (h) A recent history (in preceding 12 months) of corneal abrasions in the either eye
* (i) A recent history (in preceding 1 month) of corneal cross linking for keratoconus
* WP3:
* (a) An optometrist dispensing optician or ophthalmologist not fully registered with the General Optical Council (e.g., a pre-registration optometrist)
* (b) Hearing impairment sufficient to interfere with hearing instructions
* (c) Poor understanding of English language and/or alphabet
* (d) Any condition which, in the investigator's opinion, would conflict or otherwise prevent the participant from complying with the required procedures, schedule, or other study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with keratoconus (KC) attending Moorfields contact lens clinics
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Rigid gas permeable contact lens fit | 18 months
  The CL fit will be assessed through (i) slit lamp photography according to the standardised method proposed by Wolffsohn et al. (2013), (ii) slit lamp video of lens movement following blink in the primary position and horizontal version movements, and (iii) Anterior segment OCT MS39) (CSO Hansom Instruments, UK).

SECONDARY OUTCOMES:
The changes in contact lens fit from increased and decreased Axial Edge lift | 18 months
  Fluorescein intensity measures Wolffsohn et al. (2013) will be used to examine the predicted vs. observed alterations in contact lens fit when AEL is varied
Best corrected Visual Acuity | 18 months
  Best-corrected visual acuity with each lens design (incorporating an over-refraction where needed) will be measured using high-contrast logMAR in a forced-choice manner.
Clinician Usability Assessment | 18 Months
  Clinician Usability Assessment of topography guided virtual contact lens selection module

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom